CLINICAL TRIAL: NCT03437239
Title: Blood Flow Restriction Training After Bicep Tenodesis: A Pilot Study
Brief Title: BFR After Bicep Tenodesis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Griffin Holauchock, Orthopaedic Physician Assistant Certified Resident, Brooke Army Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: C.2018.019
Record Dates: First submitted 2018-02-13; First posted 2018-02-19 (Actual); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Shoulder Pain; Bone Mineral Density; Muscle Strength
Keywords: Bicep tenodesis
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Occlusion Training (Experimental): Patients undergoing a biceps tenodesis that are expected to begin a rehabilitation protocol with strength training by 6 weeks postoperatively for a continued 12 weeks course of 2-3 times per week of occupational therapy to include occlusion training.
  Interventions: Device: Delfi PTS II Portable Tourniquet System
- Non-occlusion Training (No Intervention): Patients undergoing a biceps tenodesis that are expected to begin a rehabilitation protocol with strength training by 6 weeks postoperatively for a continued 12 weeks course of 2-3 times per week of occupational therapy without occlusion training (standard of care).

INTERVENTIONS:
Device: Delfi PTS II Portable Tourniquet System — This is a portable tourniquet system that allows for occlusion of venous outflow without inhibiting arterial blood flow. This portable tourniquet system allows for rapid cuff inflation and deflation with a battery. The Delfi PTS is a purpose-built system that allows for precise control of pressure throughout training, despite the natural changes in muscle shape and length. The device has advanced pressure leak detection that monitors the tourniquet cuff, tubing, and connectors for air leaks and safely alerts staff to hazards or follow-up actions required. The device has visual and audio alarms for over and under pressure and elapsed time as well as a large, easily visible display of tourniquet pressure and elapsed time. The Delfi PTS II calibrates and self-tests on startup. It has a safety interlock that limits the normal maximum pressure and integrated tourniquet cuff testing as recommended in current AORN Standards and Recommended Practices
  Arms: Occlusion Training

SUMMARY:
A randomized controlled pilot study evaluating the effect of occlusion training on bone density and function of the upper extremity following a biceps tenodesis.

DETAILED DESCRIPTION:
Blood flow restriction training, resistance exercise performed with a specialized venous tourniquet, leads to beneficial changes in muscle strength at low resistance and minimal stress on the nearby joint. Early research further indicates that it improves systemic bone mineral density with change in bone turnover markers. This novel resistance training has the potential to improve muscle strength and bone density in individuals who are medically unable to perform high resistance exercises typically required to improve these attributes. Our study will examine the effect of occlusion training on bone density and function of the upper extremity following a bicep tenodesis. The primary objective of the intervention is to achieve improved bone density and accelerated recovery of upper extremity function as assessed using measures such as validated questionnaires, functional outcome testing, strength testing, and dual energy x-ray absorptiometry.

ELIGIBILITY:
Inclusion Criteria:

* Selected to undergo a unilateral bicep tenodesis
* Males and females age 18-65
* DoD beneficiaries
* Must be able to read and write in English in order to consent

Exclusion Criteria:

* Contralateral upper extremity involvement resulting in less than normal range of motion, muscle strength, or daily pain greater than 1/10.
* Rehabilitation protocol with prohibited muscle strengthening greater than 6 weeks post-operation.
* Current metallic implants that contraindicate or significantly affect the sensitivity of DEXA scan
* Current implanted defibrillator or pacemaker
* Pregnancy - per patient self-report. Due to the expected small number of pregnant individuals and resulting inability to account for its effect on resulting outcomes, these patients will not be included in this study.
* Recent history of deep vein thrombosis within the 12 months or on active treatment with anticoagulants
* Currently taking medications that are known to affect bone density to include heparin, warfarin, glucocorticoids, medroxyprogesterone acetate, cancer treatment medications, bisphosphonates or other osteoporosis treatment medications, and thyroid hormone.
* History of hyperparathyroidism
* History of upper quadrant lymph node dissection
* Patient endorsement of easy bruising
* History of an upper extremity amputation
* Active infection in the operative extremity
* Cancer (current diagnosis per medical record)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2018-02 (Estimated); Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Operative Forearm Bone Density | 24 weeks
  Bone Density will be measured using the GE Lunar Dual Energy X-ray Absorptiometry (iDXA) device maintained and operated by the Nuclear Medicine clinic at SAMMC in accordance with the International Society for Clinical Densitometry (ISCD) Best Practices for dual energy x-ray absorptiometry guidance
Total Body Bone Density | 24 weeks
  Bone Density will be measured using the GE Lunar Dual Energy X-ray Absorptiometry (iDXA) device maintained and operated by the Nuclear Medicine clinic at SAMMC in accordance with the International Society for Clinical Densitometry (ISCD) Best Practices for dual energy x-ray absorptiometry guidance
Elbow Flexion Strength | 18 weeks
  Elbow Flexion Strength will be assessed using the BTE PrimusRS dynamometer after the completion of the rehabilitation protocol, approximately 18 weeks postoperative. The patient will be seated with a lap belt to perform testing, to include isokinetic measurements of elbow flexion and forearm supination. The patient will perform 3 trials of one repetition on both the operative forearm and the contralateral arm of both elbow flexion and supination. The PrimusRS will generate a number of pounds of force used, which will be averaged for each side and used for analysis to represent strength. The BTE PrimusRS has been validated for measuring strength and used in numerous studies for various joints and movements to include elbow flexion and forearm supination
Forearm Supination Strength | 18 weeks
  Forearm Supination Strength will be assessed using the BTE PrimusRS dynamometer after the completion of the rehabilitation protocol, approximately 18 weeks postoperative. The patient will be seated with a lap belt to perform testing, to include isokinetic measurements of elbow flexion and forearm supination. The patient will perform 3 trials of one repetition on both the operative forearm and the contralateral arm of both elbow flexion and supination. The PrimusRS will generate a number of pounds of force used, which will be averaged for each side and used for analysis to represent strength. The BTE PrimusRS has been validated for measuring strength and used in numerous studies for various joints and movements to include elbow flexion and forearm supination
Grip Strength | 18 weeks.
  Grip strength will be assessed using the JAMAR Hand Dynamometer. It has been selected for use in this study as per the recommendation by the American Society for the Surgery of the Hand and American Society of Hand Therapists ASHT) as the tool of choice to measure grip strength. Studies have shown that the JAMAR dynamometer has high instrument and test-retest reliability. Grip strength will be tested according to the testing position and procedure recommended by the ASHT. The mean of three successive trials will be recorded. There are established normative data for grip strength by both age and hand dominance.

SECONDARY OUTCOMES:
Femoral Neck Bone Density | 24 weeks
  Bone Density will be measured using the GE Lunar Dual Energy X-ray Absorptiometry (iDXA) device maintained and operated by the Nuclear Medicine clinic at SAMMC in accordance with the International Society for Clinical Densitometry (ISCD) Best Practices for dual energy x-ray absorptiometry guidance
Lumbar Spine Bone Density | 24 weeks
  Bone Density will be measured using the GE Lunar Dual Energy X-ray Absorptiometry (iDXA) device maintained and operated by the Nuclear Medicine clinic at SAMMC in accordance with the International Society for Clinical Densitometry (ISCD) Best Practices for dual energy x-ray absorptiometry guidance
Pain | 24 weeks
  An 11-point verbal Numerical Rating Scale (NRS) (Appendix F) will be used to assess the subject's upper extremity pain the day of each assessment as well as during therapy sessions. The 0 to 10 NRS has been found to be valid and reliable in many patient populations including the musculoskeletal population [64] and has been recommended for inclusion in the core NIH Toolbox for use with adults
Disability of the Arm, Shoulder, and Hand | 24 weeks
  The QuickDASH consists of 11 items that measure physical function and symptoms in musculoskeletal disorders of the upper limb. The QuickDASH includes two optional scales to assess a patient's function with work activities as well as sports or playing an instrument. The QuickDASH is scored in two components: the 11-item disability section where each item is scored 1-5, and the optional work and sport/music modules. This study will only use the disability section. Respondents indicate the amount of difficulty they have performing the items (1=no difficulty, 6=unable). Scores are summed and averaged and the value is transformed to a score out of 100 by subtracting one and multiplying by 25. A higher score indicates greater disability. The QuickDASH has been validated and shown to be reliable when compared to the Disabilities of the Arm, Shoulder, and Hand
Functional Scale | 24 weeks
  The Patient Specific Functional Scale is a patient-specific outcome measure to assess functional status. The patient is asked to identify three to five activities that he or she has difficulty performing due to his or her condition. The patient then rates the amount of limitation he or she has in performing each of these activities on an 11-point scale with 0 being unable to perform the activity and 10 being able to perform the activity with no problem. An average score for the activities gives an ability score out of 10. The PSFS has been shown to be valid and responsive in the upper extremity musculoskeletal patient population

IPD SHARING:
Plan to Share IPD: No